CLINICAL TRIAL: NCT06472115
Title: A Pilot Telehealth Parent-Mediated Intervention Targeting Insistence on Sameness for Autistic Children
Brief Title: Parent-Mediated Intervention Targeting Insistence on Sameness for Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Phillips, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-73366
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Supportive Parenting for Anxious Childhood emotions (SPACE); Restricted Behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active treatment (Experimental): Eligible participants that enroll will received 16 week parent based intervention for insistence on sameness
  Interventions: Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE) for insistence on sameness (IS)

INTERVENTIONS:
Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE) for insistence on sameness (IS) — This study will examine the potential effectiveness of a virtually delivered parent-mediated intervention for insistence on sameness behaviors in autism. This includes a 16 week protocol where caregivers meet weekly for one hour with a study therapist.

SUMMARY:
This study will examine the potential effectiveness of a virtually delivered parent-mediated intervention for insistence on sameness behaviors in autism and investigate 1) whether caregivers can learn to deliver the adapted Supportive Parenting for Anxious Childhood emotions (SPACE) intervention for IS via telehealth and 2) whether children will show greater improvement in IS behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 6:0 to 10:11 years at the time of consent
* diagnosed with ASD (based on history, review of available medical records including diagnostic testing completed by psychologist)
* IQ > or = 75 (based on history, review of available medical records)
* report three or more family accommodations for insistence on sameness based on screening measures
* English-speaking parent and youth able to consistently participate in study procedures

Exclusion Criteria:

* children with significant hearing, language or motor impairment
* unstable behavioral and pharmacological treatments (e.g., anxiety medication) to treat anxiety or IS behaviors prior to two months to the start of the study and no anticipated changes in treatments during the course of the trial
* caregivers who have participated in formal SPACE training
* concurrent psychosocial treatment for anxiety or Insistence on Sameness
* children who have a history of prominent school refusal, self-harm, or suicidal ideation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parent rated Dimensional Assessment of Restricted Behavior (DARB) Scores during treatment. | Screening, Baseline, Weeks 4, 8, 12, 16 and 2 month follow up
  DARB scores measure restricted and repetitive behaviors with higher scores indicating greater intensity.
Change from baseline in clinician rated clinical global impressions scale scores during treatment. | Weeks 8, 16 and 2 month follow up
  Score Range: 1 = normal, not at all ill; 7 = among the most extremely ill patients; 1 = very much informed since the initiation of treatment; 7 = very much worse since the initiation of treatment.

SECONDARY OUTCOMES:
Change from Baseline in Parent-Rated Anxiety as captured by the Anxiety Scale for Children with Autism Spectrum Disorder (ASC-ASD). | Baseline, Week 16 and 2 month Follow up
  ASC-ASD captures anxiety with higher scores indicating greater anxiety severity across the subdomains of separation anxiety, uncertainty, performance anxiety, and anxious arousal. [Score Range: 0-72]
Change in Emotion Regulation Checklist scores during treatment | Baseline, 16 week
  The Emotion Regulation Checklist (ERC) is a 24-item measure of children's self-regulation completed by a caregiver. Items are rated along a continuum (1=rarely, 4=almost always). Higher scores on the Lability/Negativity sub scale indicate more difficulty managing and coping with emotions, while higher scores on the Emotion Regulation sub scale indicate better ability to self-regulate.
Change in Daily Living Skills Scale Scores during treatment | Baseline, 16 week, 2 month Follow up
  Higher scores indicate better ability on the DLSS. [Score Range: 0-53]
Change in Open Source - Challenging Behavior scores during treatment | Baseline, 16 weeks, 2 month Follow Up
  Higher levels indicate greater levels of challenging behavior and lower levels indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Phillips, PhD, Principal Investigator — Stanford University
Locations (1):
- Jennifer Phillips, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No